CLINICAL TRIAL: NCT05793606
Title: The Effect of Deltoid Ligament Repair in Patients With Weber B Ankle Fracture; Randomized Controlled Trial.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, Meshal Alhadhoud, Dr, Ministry of Health, Kuwait
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2156/2022
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Weber B Ankle Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deltoid repaired (Active Comparator)
  Interventions: Procedure: Deltoid ligament repair
- non-deltoid repaired (No Intervention)

INTERVENTIONS:
Procedure: Deltoid ligament repair — Surgical repair for the deltoid ligament
  Arms: Deltoid repaired

SUMMARY:
Ankle injuries are common in musculoskeletal practice with high incidence rate in physically active individuals. Ankle injuries are complex to managed and further complicated with the high recurrence rate, chronic ankle instability, and osteoarthritis (Herzog et al., 2019). The prime ankle stabilizer against valgus forces is the deltoid ligament, which is a triangle band of strong connective tissues to prevent inward ankle rotation. The deltoid ligament is vital for maintaining ankle stability against valgus forces by its deep and superficial components as it restrains eversion and external rotation of the talus on the tibia (Lee et al., 2019). The superficial components of the deltoid ligament are the tibiospring, tibionavicular, tibiocalcaneal and superficial posterior tibiotalar ligaments, while the deep components are the anterior and posterior tibiotalar ligaments. The deep components of the deltoid ligament are the main stabilizers for the ankle joint, while the superficial components have minimal stabilization role (Michelsen et al., 1996; Pankovich, 2002; Jeong et al., 2014). Retraction of the deltoid ligament could cause medial ankle instability, pain, reduce function and early osteoarthritis (Lee et al., 2019). The deltoid ligament is essential for normal functioning of the foot and ankle and to maintain the normal kinematics of the talocrural kinematics. Dodd, Halai and Buckely (2022) discussed based on Ramsey and Hamilton's (1976) and Lubbeke et al..'s (2012) studies that a one mm lateral shift of the talus reduces the contact area of the tibiotalar up to 42%, and medial-sided injuries including an injury to the deltoid ligament would lead to long-term arthritis (Ramsey and Hamilton, 1976; Lubbeke et al., 2012; Dodd, Halai amd Buckley, 2022). More importantly, the deltoid ligament frequently raptures in association with ankle fractures (Wang et al., 2020). However, a recent systematic review stated that there is no consensus regarding deltoid ligament repair and its associated effectiveness and complications (Dodd, Halai and Buckely, 2022). Moreover, no study has explored the long-term effect of deltoid ligament repair in reducing post-traumatic ankle instability and osteoarthritis in patients with weber B fibula fractures. Therefore, the aim of the study is to determine the effect of deltoid ligament repair in patient with Weber B fibular fracture using randomized controlled trial design and two years follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male subjects.
2. Age 18-55 years.
3. Diagnosed with isolated weber B fibula facture with deltoid ligament injury confirm with radiography, MRI and CT scan. CT scan will be used to see the rotational element of the talus in the axial cuts and MRI to confirm the superficial ligament rupture.
4. Assigned for ORIF for the fibula.
5. One surgeon (MA) will perform the surgical intervention

Exclusion Criteria:

1. Patient with open fractures and syndesmotic injury
2. Previous ankle injury.
3. Multiple trauma of the lower extremities.
4. Rheumatoid arthritis or other chronic inflammatory condition.
5. Previous history of ankle instability
6. Ankle osteoarthritis
7. No osteochondral lesion
8. BMI > 35

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Ankle instability measured with the Cumberland Ankle Instability Tool (CAIT) | two years

SECONDARY OUTCOMES:
• Foot and Ankle Ability Measure | two years
• Global Rating of Function | two years
• AOFAS | two years
SF-12 | two years
VAS | two years
• EQE5 | two years

IPD SHARING:
Plan to Share IPD: Undecided